CLINICAL TRIAL: NCT07134868
Title: The Diagnostic Efficacy of Thiol-Disulfide Homeostasis in Sepsis Patients
Brief Title: Sepsis and Thiol-Disulfide Balance in Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Mehmet Alaçam, MD, Medicine Doctor, Sakarya University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SAU-ED-MA-01
Record Dates: First submitted 2024-06-27; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Sepsis; Oxidative Stress
Keywords: Diagnostic efficacy; Sepsis; Oxidative Stress; Emergency Department; Thiol- Disulfide Homeostasis
MeSH Terms: conditions — Sepsis; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sepsis Group (Active Comparator): Consisted of patients diagnosed with sepsis (defined as those presenting to the emergency department with suspected infection and scoring two or higher on the quick Sequential Organ Failure Assessment scoring system according to the Sepsis-3 guidelines) and who agreed to participate in the study.
  Interventions: Diagnostic Test: Thiol- Disulfide Blood Sample Measurement
- Control Group (No Intervention): Comprised of healthy volunteers who presented to the emergency department for any reason and agreed to participate in the study.

INTERVENTIONS:
Diagnostic Test: Thiol- Disulfide Blood Sample Measurement — Measurement of thiol-disulfide homeostasis parameters and inflammatory markers from serum samples.
  Arms: Sepsis Group

SUMMARY:
The aim of this study was to determine the effectiveness of thiol-disulfide homeostasis in predicting diagnosis and mortality in sepsis patients, and to compare it with other inflammatory markers.

DETAILED DESCRIPTION:
Sepsis is a serious illness with high mortality rates triggered by infection-associated pathogenesis involving oxidative stress dysfunction. This study aims to elucidate the diagnostic efficacy of changes in thiol-disulfide homeostasis, its predictive role in mortality, relationship with other inflammatory parameters in sepsis patients in emergency department.

In prospective, randomized controlled study, 50 patients diagnosed with sepsis according to the Sepsis-3 guidelines who presented emergency department were compared with a control group of 50 healthy volunteers. Thiol-disulfide homeostasis parameters, including total thiol, native thiol, disulfide levels, reduced thiol, oxidized thiol, and thiol oxidation-reduction ratios, were examined. Additionally, inflammatory blood parameters (C-reactive protein, procalcitonin, lactate) and mortality durations were compared with thiol-disulfide homeostasis.

The objective of this study was to examine the effectiveness of thiol-disulfide homeostasis in forecasting diagnosis and mortality in sepsis patients, and to compare it against other inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and above who met the diagnostic criteria were included in the study

Exclusion Criteria:

* Who did not meet the criteria for sepsis diagnosis according to the quick Sequential Organ Failure Assessment score
* Individuals with malignancy, acute coronary syndrome, acute cerebrovascular event, acute/chronic kidney/liver failure, rheumatologic diseases, febrile neutropenia, immunosuppressive disorders, corticosteroid use, and those
* Individuals with a history of antibiotic use within the last week

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Diagnostic value of serum thiol-disulfide homeostasis parameters in sepsis | 2 monhts
  Measurement of serum total thiol, native thiol, disulfide, reduced thiol, and oxidized thiol levels in patients with sepsis and healthy controls at the time of admission, and comparison between groups to evaluate diagnostic performance.

SECONDARY OUTCOMES:
General Characteristics of All Participants | 1 week
  Demographic data (age, gender, body mass index) were recorded.
Correlation of inflammatory and biochemical markers with thiol-disulfide homeostasis in sepsis | 10 days
  Initial blood samples collected from sepsis patients were analyzed to measure total thiol, native thiol, disulfide, reduced thiol, and oxidized thiol levels. These thiol-disulfide homeostasis parameters were then compared and correlated with standard laboratory inflammatory markers, including C-reactive protein (CRP), procalcitonin, and lactate, to evaluate their relationships.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Alacam, M.D., Principal Investigator — Sakarya University
Locations (1):
- Sakarya University, Sakarya, Adapazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No